CLINICAL TRIAL: NCT02190331
Title: The Effects of Training and Detraining After an 8 Month Resistance and Stretching Training Program on Forward Head and Protracted Shoulder Postures in Adolescents
Brief Title: Effects of a Resistance and Stretching Training Program on Forward Head and Protracted Shoulder Posture Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Rodrigo Ruivo, Mr Rodrigo Ruivo, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/77633/2011
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Posture Disorders in Children
Keywords: Detraining; Neck; Exercise; Posture; Rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional program (Experimental): The training protocol is constituted by 4 strengthening exercises (Side Lying External Rotation, Prone Horizontal Abduction with External Rotation, Y to I exercise and Chin Tuck) and 3 stretching exercises(one- Sided Unilateral Self Stretch Exercise, one-sided Unilateral Self Stretch Exercise, Static Sternocleidomastoid Stretch and Static Levator Scapulae Stretch
  Interventions: Other: Interventional program postural correction training
- Control group (Active Comparator): The control group will only participate in the Physical Education classes
  Interventions: Other: Control Group physical education classes

INTERVENTIONS:
Other: Interventional program postural correction training — The postural correction training program was applied in the last 15-20 minutes of each PE class, twice a week, with the supervision and help of the PE teacher.
  Arms: Interventional program
Other: Control Group physical education classes — Only performed the physical education classes
  Arms: Control group

SUMMARY:
* To evaluate the effects of a 32-weeks resistance and stretching training program applied in Physical Education classes on forward head and protracted shoulder Portuguese adolescents (15-17 years old).
* To evaluate on adolescents submitted to strength and stretching exercises the effects of a 16-week detraining period after the end of the intervention protocol.

DETAILED DESCRIPTION:
A prospective, randomized and controlled study will be conducted over a 12 month period, with adolescents of two public secondary schools, in Lisbon.

At the beginning, a total of 275 adolescent students aged 15-17 years old will be evaluated with photogrammetry. The students will be screened by measuring the cervical (CV) and shoulder (SH) angle with photogrammetry. If the CV and SH angle were less than 50º and 52º respectively, the adolescent was considered to have forward head posture (FHP) and protracted shoulder (PS) and was selected to the study.

Participants will be excluded if their CV and SH angle was equal or higher than 50º and 52º respectively, if they had visual deficits, diagnosed balance disorders, musculoskeletal pathologies, such as a history of shoulder surgery, cervical or thoracic fracture, were non-ambulatory, displayed functional or structural scoliosis, or had excessive thoracic kyphosis.

After these the eligible students will be randomly assigned to the control or interventional group. The intervention group will begin a 32-week stretching and strengthening program to be performed in the last part of the Physical Education (PE) classes. The control group will only participate in the PE classes. Since the 32th week until the 48th week the experimental group will not follow the interventional training program and both groups will only participate in PE classes.

The program will be constituted by four strengthening exercises and three stretching exercises and is designed based on the assumption that the use of therapeutic exercise is effective in the correction of specific neck and shoulder postures. The training exercise protocol will be designed for the correction of the FHP and PS, targeting to the selective activation of lower trapezius, middle trapezius and rhomboids, to the lengthening of the pectoralis major, pectoralis minor and sternocleidomastoid and to the improvement of the deep cervical flexor function This program is going to be applied in the last 15-20 minutes of each PE class, twice a week, with the supervision and help of the PE teacher.

The postural assessment of the groups will be performed in the beginning and after 36 and 48-weeks intervention period.

ELIGIBILITY:
Inclusion Criteria:

adolescents with 15-17 years old with cervical angle lower than 50º and the shoulder angle lower than 52º

Exclusion Criteria:

Participants were excluded if their CV and SH angle was equal or higher than 50º and 52º respectively, if they had visual deficits, diagnosed balance disorders, musculoskeletal pathologies, such as a history of shoulder surgery, cervical or thoracic fracture, were non-ambulatory, displayed functional or structural scoliosis, or had excessive thoracic kyphosis.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
change in postural angles (cervical and shoulder angle) | 36 and 48 weeks
  We will assess the Cervical angle - the angle formed at the intersection of a horizontal line through the spinous process of C7 and a line to the tragus of the ear and the shoulder angle - The angle formed at the intersection of the line between the midpoint of the humerus and the spinous process of C7 and the horizontal line through the midpoint of the humerus.

SECONDARY OUTCOMES:
the American Shoulder and Elbow Surgeons Standardized questionnaire | 36 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruivo, Master, Principal Investigator — University of Lisbon
Locations (1):
- Technical University of Lisbon, Lisbon, Cruz Quebrada-Dafundo, Portugal

REFERENCES:
- [Derived] Ruivo RM, Pezarat-Correia P, Carita AI. Effects of a Resistance and Stretching Training Program on Forward Head and Protracted Shoulder Posture in Adolescents. J Manipulative Physiol Ther. 2017 Jan;40(1):1-10. doi: 10.1016/j.jmpt.2016.10.005. Epub 2016 Nov 11. PMID 27842938
- [Derived] Ruivo RM, Carita AI, Pezarat-Correia P. The effects of training and detraining after an 8 month resistance and stretching training program on forward head and protracted shoulder postures in adolescents: Randomised controlled study. Man Ther. 2016 Feb;21:76-82. doi: 10.1016/j.math.2015.05.001. Epub 2015 May 13. PMID 26028408